CLINICAL TRIAL: NCT01581099
Title: Effect of Bariatric Surgery "Digestive Adaptations III" on Clinical, Laboratory and Cardiovascular Risk Factors
Brief Title: Effect of Bariatric Surgery "Digestive Adaptations III" on Cardiovascular Risk
Acronym: ADIII
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Bruno Caramelli, Director, Interdisciplinary Medicine in Cardiology Unit, Heart Institute, University of Sao Paulo
Other Study IDs: USP - 0355/11
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus; Metabolic Syndrome; Obesity; Atherosclerosis
Keywords: Atherosclerosis; Cardiovascular risk factors; Calorie restriction; Bariatric Surgery
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Syndrome; Obesity; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples will be retained for future exams.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Clinical treatment: Diabetic individuals refractory to medical treatment kept under clinical treatment guidelines and lifestyle
- Surgery: Diabetic individuals refractory to conservative clinical treatment subject to Digestive Adaptations III Surgery.
  Interventions: Procedure: Digestive Adaptations III surgery
- Control: Healthy individuals (normal weight and no cardiovascular risk factors) will be used to evaluate the behavior incretin hormones in healthy individuals, serving as a benchmark to analyze the results obtained in other groups.

INTERVENTIONS:
Procedure: Digestive Adaptations III surgery
  Other Names: Sleeve gastrectomy with transit bipartition
  Groups: Surgery

SUMMARY:
Introduction- Primary prevention is the main strategy to control the global burden of cardiovascular disease. In clinical practice, food restriction represents a valuable preventive resource. However, low adhesion rates and diet abandonment are considered important obstacles in treatment. Considering the discovery of new markers and mechanisms that relate food restriction and to all other cardiovascular risk factors, it is possible and necessary to seek for efficient alternatives to increase adherence and effectiveness of the preventive dietetic treatment. Surgical procedures can be used as a mechanism to promote food restriction. The bariatric surgery have gained importance not only for its potential application in obesity treatment but also in the control of cardiovascular risk factors refractory to medical treatment. Among bariatric operations, there is a group called digestive adaptations III that has specific characteristics.This surgical intervention modifies intestinal tract by reducing gastric volume and performing an anastomosis between ileum and stomach, creating a bipartition in the gut. This structural modification promotes satiety and increased insulin sensitivity more intensely than other surgical strategies. The effects of Digestive Adaptation III surgery on cardiovascular risk factors and on markers related to the development of atherosclerosis are not yet established.

Objectives - To investigate the effect of Digestive Adaptation III surgery on clinical and laboratory parameters and cardiovascular risk factors.

Methods - Twenty diabetics volunteers refractory to medical treatment and who have abdominal obesity will be included in the study. Of this group, half will be randomly selected to perform the Digestive Adaptations III surgery. All participants will undergo clinical and biochemical tests on the same occasions, up to thirty days before surgery, three twenty-four months after surgery. On these occasions besides the lipid profile and glucose, we will determine incretin hormones, adipokines and assess the amount of epicardial fat.

ELIGIBILITY:
Inclusion Criteria:

* Men.
* Adults (raging from 18 to 65 years).
* Ability to understand the procedure, risks and alternatives.
* Patients with BMI > 28 Kg/m2 and < 35 Kg/m2 presenting type 2 diabetes diagnosed for more than two years and less than 10 years.
* Glycated hemoglobin> 8% despite dietary and medical treatment that already includes the use of exogenous insulin
* Waist circumference > 102 cm.

Exclusion Criteria:

* Chronic diseases not related to severe obesity.
* Pregnancy.
* Peptide C <1.5 ng / mL or a positive anti-islet antibodies, anti-GAD or anti-ICA512.
* Previous cancer, unless deemed cured (after 5 years of treatment, at least)
* Acute infection or chronic relevant.
* Alcohol addiction.
* Tobacco use.
* Drug addiction, except those recovered for more than three years.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will be selected in a primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2016-03 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Improvement in Metabolic Profile | two years
  Modification in variables linked to cardiovascular diseases leading to an estimated reduction in cardiovascular risk.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Caramelli, Ph.D., Study Chair — University of Sao Paulo; Fernanda R Azevedo, Nutr, Principal Investigator — University of Sao Paulo
Locations (1):
- Heart Institute - University of São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Azevedo FR, Santoro S, Correa-Giannella ML, Toyoshima MT, Giannella-Neto D, Calderaro D, Gualandro DM, Yu PC, Caramelli B. A Prospective Randomized Controlled Trial of the Metabolic Effects of Sleeve Gastrectomy with Transit Bipartition. Obes Surg. 2018 Oct;28(10):3012-3019. doi: 10.1007/s11695-018-3239-3. PMID 29704228